CLINICAL TRIAL: NCT02651389
Title: Evaluation de la Performance d'Une Nouvelle Plateforme de Tests de dépistage Orthoptique numériques
Brief Title: Evaluation of Tests Performance on a New Digital Orthoptic Platform
Acronym: ESPPADON
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RB 15.087 - ESPPADON
Record Dates: First submitted 2015-12-29; First posted 2016-01-11 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Binocular Vision Disorder; Visual Impairment
Keywords: Digital Orthoptic Platform; Vision test
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical trials aims to evaluate Tests Performance on a New Digital Orthoptic Platform.

DETAILED DESCRIPTION:
The demography of ophthalmologists is becoming weaker, many tasks are now performed by orthoptists. To optimize the achievement of orthoptic exams and thus make reliable screening in a shorter time, digital tools are developed. They attempt to renew the orthoptic screening equipment that is still made up of numerous tests, often with old designs that must be handled and adapted to each patient which constitutes a significant loss of time.

It therefore appeared necessary for us to develop a platform of digital tools that integrates major tests used for diagnostic purposes, especially a visual acuity test, a stereoscopic vision test, a fusion test and a digital synoptophore enabling a detailed analysis of disorders of binocular vision.

The purpose of the study is to evaluate this new tool, avoiding the mobilization of patients , and quantify whether this platform is precise, reliable, fast, comfortable and allow the realization of a safe examination for the patient and for orthoptics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with less than or equal to 16 ocular deviation prism diopters, without or with slight amblyopia (maximum difference of 2 logarithmic visual acuity lines) and performing an orthoptic exam at ophthalmology department of Brest University Hospital.

Exclusion Criteria:

* monophthalmic
* Medium and deep amblyopic patients
* Patients with not normal ocular motility
* Patient who underwent surgery at the head and neck during the previous three months
* Children under 7 years old.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People performing an orthoptic exam at ophthalmology department of Brest University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Correlation of Ocular Convergence as Measured by the Two Machines | through study completion, an average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Cochener, Pr, Principal Investigator — University Hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No